CLINICAL TRIAL: NCT07182175
Title: Dynamic Monitoring and Comparative Study of Perioperative Cardiac Injury in Patients With Functional Adrenal Tumors
Brief Title: Comparative Study of Perioperative Cardiac Injury in Patients With Functional Adrenal Tumors
Status: Enrolling by invitation | Type: Observational
Sponsor: Peking University First Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2024yan411-002
Record Dates: First submitted 2025-09-11; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Primary Aldosteronism; Adrenal Tumor; Cushing s Syndrome; Pheochromocytoma/Paraganglioma (PPGL)
MeSH Terms: conditions — Hyperaldosteronism; Adrenal Gland Neoplasms; Pheochromocytoma; Paraganglioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 48 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- primary aldosteronism
- Cushing s Syndrome
- Pheochromocytoma/Paraganglioma (PPGL)

SUMMARY:
The main goal of this study is to follow patients with functional adrenal tumors during the time before and after their surgery.

The main questions it aims to answer are:

* What heart and blood pressure changes do patients with different types of adrenal tumors have before surgery?
* What factors affect how the heart and blood pressure recover after surgery?
* Do the heart and blood pressure conditions before surgery influence recovery and the risk of heart or brain problems after surgery?

Patients will have heart ultrasound checks and health monitoring before and after surgery. The results will help doctors choose the right medicines before surgery, better understand possible risks during the operation, and make safer treatment plans for patients with functional adrenal tumors.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed in the Department of Urology, Peking University First Hospital with pheochromocytoma and paraganglioma (PPGL), primary aldosteronism (PA), or Cushing syndrome (CS);
* Written informed consent obtained.

Exclusion Criteria:

* Patients with PPGL, PA, or CS who receive medication or conservative treatment and are not eligible for surgical resection;
* Patients with communication disorders or severe physical impairments such as aphasia, or visual/hearing disabilities;
* Patients with severe mental illness who cannot cooperate with the study;
* Pregnant women or patients otherwise deemed unsuitable for participation by the investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients with functional adrenal tumors who are hospitalized and/or seen in the outpatient clinic of the Department of Urology at Peking University First Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-09-19 (Actual); Primary Completion 2024-11-17 (Actual); Study Completion 2026-05-29 (Estimated)

PRIMARY OUTCOMES:
Recovery of cardiac function after adrenal surgery | from enrollment to 4,24,48 weeks after surgery
  global longitudinal stress

SECONDARY OUTCOMES:
Recovery of blood pressure after adrenal surgery | from enrollment to 4,24,48 weeks after surgery
  Decrease in 24h average blood pressure

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No
Data cannot be shared, because data from this study may contain potentially or sensitive patient information.